CLINICAL TRIAL: NCT06458959
Title: Patient-Reported Outcomes Plus Care Planning Applications for Strengthening Participation on Early Intervention Care Teams
Brief Title: Exploratory Trial of a Pediatric Web-Based Care Planning Guide
Acronym: PROSPECT+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Rocky Mountain Human Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-0908
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Developmental Disabilities; Developmental Delay
Keywords: early intervention; participation; childhood disability; environment; families; family-centered care
MeSH Terms: conditions — Developmental Disabilities; Learning Disabilities

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: cluster randomization at the service coordinator level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEM+ (Experimental)
  Interventions: Behavioral: PEM+
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: PEM+ — The Young Children's Participation in Environment Measure (YC-PEM), an evidence-based and promising electronic patient-reported outcome (e-PRO) when combined with the Participation and Environment Measure Plus (PEM+) care planning application that yields a summary report and is paired with a program-specific decision-support tool, may support family engaged Early Intervention (EI) service plan development. Intervention group caregivers will complete the YC-PEM e-PRO and PEM+ intervention before their child's annual review of progress. The online summary report will be combined with a program-specific decision-support tool to guide EI service plan development.
  Arms: PEM+

SUMMARY:
Infants and toddlers with developmental disabilities or delays use early intervention (EI) for rehabilitation services. Yet, poor quality of EI services is pervasive, particularly for racially and ethnically diverse and socially disadvantaged families. A key lever to improve EI quality is family-centered care, an evidence-based approach that is grounded in family engagement for shared decision-making. This project is motivated by the need to give families a smart and connected option for engaging in the design of the EI service plan for their child. This project upgrades and tests an evidence-based and innovative electronic solution that helps families to organize and share their priorities for change and ideas for goal attainment with professionals, so as to ensure fit of the service plan with their needs.

DETAILED DESCRIPTION:
Infants and toddlers with developmental disabilities or delays use early intervention (EI) for rehabilitation services. Yet, poor quality of EI services is pervasive, particularly for racially and ethnically diverse and socially disadvantaged families. A key lever to improve EI quality is family-centered care, an evidence-based approach that is grounded in family engagement for shared decision-making.

This project further develops and evaluates the Participation and Environment Measure (PEM), an electronic option for family-centered EI service design that has two parts: 1) an evidence-based and promising electronic patient-reported outcome (e-PRO) assessment called the Young Children's Participation and Environment Measure (YC-PEM), and 2) a prototypic goal setting application called Participation and and Environment Measure Plus (PEM+). This project builds on published evidence for its feasibility, acceptability, and preliminary effectiveness of the YC-PEM e-PRO, when paired with a program-specific decision-support tool, on EI service quality. EI stakeholder perspectives on salient supports, barriers, and strategies signal its viability for broader early intervention service system implementation. One important optimization involves expanding its reach to historically minoritized families.

This project will be accomplished in 3 aims: 1. The PEM assessment and intervention content will be culturally adapted to amplify the assessment and consideration of racial climate on young children's participation in activities during the design of an EI service plan (i.e., make content more relevant for racially and ethnically diverse EI families). 2. Artificial intelligence (AI) will be applied to personalize the user experience of the PEM intervention to a broader range of EI enrolled families (i.e., leverage the power of natural language processing as a form of AI, to individualize the PEM intervention to caregivers in two ways). 3. The team will evaluate the effectiveness of the upgraded PEM electronic option to improve caregiver perceptions of family-centered service quality, improve parent engagement in EI service plan implementation, and increase the proportion of participation-focused EI service plans. EI family and provider perspectives will be obtained on supports, barriers, and strategies to its broader implementation in the early intervention service system.

ELIGIBILITY:
Inclusion Criteria:

* read, write, and speak English,
* have internet and telephone access
* identify as a parent/legal guardian of a child enrolled in EI for 3+ months

Exclusion Criteria:

* do not read, write, and speak English
* do not have internet and phone access
* do not identify as a parent/legal guardian of a child enrolled in EI for 3+ months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Rehabilitation Intervention Measure of Engagement - Parent version (PRIME-P) | baseline, 4 weeks, 3 months
  11-item self-report measure that asks parents what they thought, how they felt, and what they did during their child's therapy session and how the session has affected their overall feelings about the intervention process.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No